CLINICAL TRIAL: NCT04647422
Title: Investigation of Social Cognition and Executive Functions as Cognitive Vulnerability Markers for the Development and Maintenance of Alcohol Use Disorders - a Transverse Study Design
Brief Title: Social Cognition and Executive Functions in Alcohol Use Disorders - Transverse Study
Acronym: COSEFEX-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO20089
Record Dates: First submitted 2020-09-16; First posted 2020-11-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol use disorder; high-risk individuals; executive functions; social cognition; endophenotypes; neuropsychology
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AUD patients (Experimental): Alcohol Use Disorder patients
  Interventions: Behavioral: Analysis of executive functioning and of social cognition processes
- AUD controls (Experimental): Healthy control participants matched to group 1
  Interventions: Behavioral: Analysis of executive functioning and of social cognition processes
- First-degree relatives (Experimental): Healthy first-degree relatives of AUD patients
  Interventions: Behavioral: Analysis of executive functioning and of social cognition processes
- First-degree controls (Experimental): Healthy control participants matched to group 3
  Interventions: Behavioral: Analysis of executive functioning and of social cognition processes

INTERVENTIONS:
Behavioral: Analysis of executive functioning and of social cognition processes — Investigation of executive and social cognition processes using a comprehensive, neuropsychological assessment, An Eye tracking investigation and Task-based MRI exams.
  * Evaluation of addictive, psychiatric and neurological comorbidities.
  * Neuropsychological assessment establishing the participants' cognitive profiles of executive functions and of social cognition
  * An Eye tracking investigation aiming at a better understanding of participants' emotional processing
  * Task-based MRI exams identifying participants' neuroanatomical and neurofunctional correlates of executive functions and of social cognition processes

SUMMARY:
Over the past few years, researchers and clinicians have stressed the major role of executive and social cognition impairments in the development and the maintenance of Alcohol Use Disorders (AUD).

Executive functions are defined as functions for behavioral control that help us to adjust the investigator's behavior in a flexible way in non-familiar, non-routine situations. Executive functions encompass different cognitive processes, such as inhibition, mental flexibility, updating, planification, abstraction, rule deduction or organization. Studies comparing AUD patients to healthy controls have shown that AUD usually is associated with a large range of deficits. More recently studies have also emphasized a weakness of executive functioning among healthy participants with a positive family history of AUD.

Social cognition refers to all cognitive processes that enable us to communicate and to interact with social environment in an appropriate manner. Among the most common social cognition sub-components are theory of mind (defined as the capacity to understand other people's mental states as for instance beliefs and desires), empathy, and emotion recognition. Emotional and interpersonal difficulties have a high prevalence in AUD and chronic alcohol consumption is often linked to social conflicts, misunderstandings, a lack of social support and isolation. Indeed, AUD patients have difficulties in understanding their own mental states and emotions as well as those of their social environment.

Few studies have investigated the interdependency between these cognitive impairments in AUD while a better understanding of the link between executive functions and social cognition seems crucial in order to better characterize the nature of AUD patients' deficits and thus their caring.

DETAILED DESCRIPTION:
The aim of the study is to describe cognitive processes (theory of mind, empathy, and emotion recognition) and executive functions (inhibition, mental flexibility) in patients with AUD and first degree relatives of patients with an AUD.

ELIGIBILITY:
1. AUD patients

   Inclusion criteria:
   * Patients between 18 and 60 years old, men or women, following AUD treatment
   * Having a diagnosis of alcohol use disorder according to DSM-5 criteria
   * Patients withdrawn of alcohol for at least 15 days
   * Patients being a native French speaker
   * Patients enrolled in the national healthcare insurance program
   * Patients consenting to participate to the study

   exclusion criteria:
   * A diagnosis of schizophrenia, of any other chronic psychotic state, or of bipolar disorder according to DSM-5 criteria
   * The presence of a current depressive episode as defined by DSM-5 criteria
   * The presence of another substance use disorder during the six months preceding the study, except for tobacco dependence.
   * The presence of any intellectual disability, of pervasive developmental disorders or learning difficulties (especially of dysphasia and dyspraxia)
   * The presence of any neurological disorder or any other disorder affecting the central nervous system including Korsakoff syndrome or Wernicke's encephalopathy
   * Having any uncorrected auditory or visual deficits
2. First-degree relatives of AUD patients

   Inclusion criteria:
   * Participants between 18 and 60 years old, men or women
   * Current and past absence of any alcohol use disorder or any other substance use disorder as defined by DSM-5 diagnostic criteria
   * Participants having at least one first-degree relative presenting an alcohol use disorder (father or sibling)
   * Participants being a native French speaker
   * Participants enrolled in the national healthcare insurance program
   * Participants consenting to participate to the study

   exclusion criteria:
   * The presence of any alcohol use disorder or any other substance use disorder as defined by DSM-5 diagnostic criteria, except for tobacco dependence
   * A diagnosis of schizophrenia, of any other chronic psychotic state, or of bipolar disorder according to DSM-5 criteria
   * The presence of a current depressive episode as defined by DSM-5 criteria
   * The presence of any alcohol use disorder in the participant's biological mother in order to exclude fetal alcohol spectrum disorders due to prenatal alcohol intoxication
   * The presence of any intellectual disability, of pervasive developmental disorders or learning difficulties (especially of dysphasia and dyspraxia)
   * The presence of any neurological disorder or any other disorder affecting the central nervous system
   * Participants having any uncorrected auditory or visual deficits
3. Healthy control participants (the inclusion and non-inclusion criteria of investigation groups 2 and 4 are identical):

Inclusion criteria:

* Participants between 18 and 60 years old, men or women
* Current and past absence of any alcohol use disorder or any other substance use disorder as defined by DSM-5 diagnostic criteria
* Participants being a native French speaker
* Participants enrolled in the national healthcare insurance program
* Participants consenting to participate to the study

exclusion criteria:

* The presence of any alcohol use disorder or any other substance use disorder as defined by DSM-5 diagnostic criteria, except for tobacco dependence
* A diagnosis of schizophrenia, of any other chronic psychotic state, or of bipolar disorder according to DSM-5 criteria
* The presence of a current depressive episode as defined by DSM-5 criteria
* Having any first-degree relative with alcohol use disorder (parents, siblings, children) according to DSM-5 diagnostic criteria
* The presence of any intellectual disability, of pervasive developmental disorders or learning difficulties (especially of dysphasia and dyspraxia)
* The presence of any neurological disorder or any other disorder affecting the central nervous system
* Participants having any uncorrected auditory or visual deficits

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Executive functions: mental flexibility performances and processing speed | Day 0
  Evaluated through the Trail Making Test (TMT parts A and B). In part A the participant must connect as quick as possible all the numbers on a sheet of paper in ascending order (1-25). In part B the participant is asked to connect all the numbers in ascending order (1-13) and all the letters according to their alphabetical order (A-L) whilst alternating between numbers and letters and without lifting the pencil. For both parts is reported the time necessary for task completion in seconds.
  (Reitan RM, Wolfson D (1985) The Halstead-Reitan Neuropsychological Test Battery. Neuropsychology Press, Tucson, AZ.)
Executive functions: mental flexibility performances | Day 0
  Evaluated through the Plus-Minus test. In this test, the participant is presented with three lists of 30 two-digit numbers. At first, the participant is asked to add three to all the numbers of a first list (+3). He must then subtract three from all the numbers of a second list (-3) and finally he must alternate between addition and subtraction when presented with a third list (+3/-3). Are measured the completion times for the three lists and participant's error rate.
  (Miyake A, Friedman NP, Emerson MJ, Witzki AH, Howerter A, Wager TD (2000) The unity and diversity of executive functions and their contributions to complex "Frontal Lobe" tasks: a latent variable analysis. Cognitive Psychology 41, 49-100.)
Executive functions: prepotent response inhibition | Day 0
  Evaluated through the Stroop test. The participant is shown three different slides with 100 items for 45s each. On the first slide are written color words (Color-word congruent condition) that the participant must read as quickly as possible. On the second slide are shown color patches (Color congruent condition) that the participants must name as quickly as possible. Finally, in the third condition, the participant is shown color words written in different colors and must try to name the color of the ink of the word without reading it (Interference condition). Are collected the completion times for the tree slides as well as self-corrected and uncorrected errors.
  (Golden C.J (1976) Identification of brain disorders by the Stroop color and word test. Journal of Clinical Psychology 32, 654-658)
Executive functions: inhibition of an ongoing motor response | Day 0
  Evaluated through the Stop signal task. The participant is presented with a series of photographs showing human faces and is instructed to categorize the photographs according to gender (Go trials). From time to time a red circle appears around the face after a variable time interval and the participant must then withhold his response (Stop trials). Are measured the response time on Go trials, the number and type of errors and the Stop Signal Reaction Time (SSRT).
  (Verbruggen F., & Logan G.D. (2008) Response inhibition in the stop-signal paradigm. Trends in cognitive sciences 12, 418-424.)
Social cognition: facial emotion recognition | Day 0
  Evaluated through a test of facial emotion recognition (TREF). The participant is shown 54 photographs depicting 6 different emotions of variable intensity (joy, anger, sadness, disgust, contempt, fear) for which he must choose the corresponding emotion label. Are measured participant's response times, the number of correct responses (score out of 54) and type of errors.
  (Gaudelus, B., Virgile, J., Peyroux, E., b, Leleu, A., c, Baudouin J.Y., Franck N. (2015). Mesure du déficit de reconnaissance des émotions faciales dans la schizophrénie. Étude préliminaire du test de reconnaissance des émotions faciales (TREF). L'encéphale 41(3), 251-259.)
Social cognition: cognitive and affective theory of mind | Day 0
  Evaluated through The Movie of Assessment for Social Cognition (MASC). The participant is shown a movie of approximately 15 minutes displaying people interacting with each other. From time to time, the movie is stopped, and the participant must answer different questions relating to the thoughts and feelings of the characters. Are measured the number of correct responses out of 45.
  (Dziobek I, Fleck S, Kalbe E, Rogers K, Hassenstab J, Brand M, Kessler J, Woike JK, Wolf OT, Convit A.J (2006). Journal of Autism and Developmental Disorders 36(5), 623-36.)

SECONDARY OUTCOMES:
Duration of ocular fixations | Day 0
  The mean duration of fixations will be evaluated using eye tracking. The participant is shown photographs of primary emotions and during the presentation are recorded his eye movements.
Number of ocular saccades | Day 0
  The number of saccades will be evaluated using eye tracking. The participant is shown photographs of primary emotions and during the presentation are recorded his eye movements.
Localization of the first ocular fixation | Day 0
  The localization of the first fixation will be evaluated using eye tracking. The participant is shown photographs of primary emotions and during the presentation are recorded his eye movements.
fMRI behavioral responses during a cognitive and affective theory of mind task | Day 0
  During the task will be recorded the participant's behavioral performance (number of correct responses).
fMRI activations during a cognitive and affective theory of mind task | Day 0
  Brain regions significantly activated during the task will be recorded as shown by the variations in the BOLD signal (whole brain analysis).

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Result] Schmid F, Henry A, Benzerouk F, Barriere S, Gondrexon J, Kaladjian A, Gierski F. Patterns of executive functions and theory of mind in adults with a family history of alcohol use disorder: Combined group and single-case analyses. Alcohol Clin Exp Res (Hoboken). 2024 Feb;48(2):362-374. doi: 10.1111/acer.15238. Epub 2024 Jan 20. PMID 38243915